CLINICAL TRIAL: NCT06078176
Title: Electrical Rectal Stimulation to Promote Bowel Emptying After Spinal Cord Injury
Brief Title: Stimulation for Bowel Emptying
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4529-R
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Neurogenic Bowel Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bowel emptying (Experimental): Study participants will act as their own controls, first providing data using their usual digital rectal stimulation intervention for bowel care, then providing data using electrical stimulation for bowel care.
  Interventions: Other: Electrical Rectal Stimulation

INTERVENTIONS:
Other: Electrical Rectal Stimulation — Electrical stimulation of the rectum will be applied to activate sensory afferent neurons of the rectum and evoke a recto-colonic reflex to improve colonic motility and facilitate bowel emptying. This intervention will compared to individuals' usual mechanical intervention of digital rectal stimulation.

SUMMARY:
The investigators are testing the effect of electrical stimulation of the rectum on colonic motility. Most individuals with spinal cord injury develop neurogenic bowel dysfunction, which includes slowed colonic motility, which means that stools take longer than normal to pass through the colon. This slowed movement may result in chronic constipation and difficulty emptying the bowels. Individuals typically (without or without caregiver assistance) insert a gloved finger into the rectum and gently stretch it to improve colonic motility for a brief period to empty the bowels. The investigators hypothesize that electrically stimulating the rectum, instead of mechanically stretching it, will produce the same beneficial effect of improving colonic motility. Therefore, this study will compare the two methods. If electrical stimulation effectively improves colonic motility, then the investigator shall develop the approach as a therapeutic intervention in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Suprasacral spinal cord injury
* Diagnosed neurogenic bowel dysfunction and using digital rectal stimulation
* Bowel routine requires at least 30 minutes or at least 3 cycles of digital rectal stimulation
* Neurologically stable
* At least 18 years old
* At least 12 months post neurological injury or disease diagnosis

Exclusion Criteria:

* Active sepsis
* Open pressure sores on or around pelvis
* Significant colon trauma or colostomy
* Crohn's disease
* Colonic obstruction or gastrointestinal surgery within last 3 months
* Significant history of autonomic dysreflexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time required to complete bowel emptying | 12 weeks
  Two interventions will be tested, including the clinical standard of digital rectal stimulation and a novel approach using electrical stimulation of rectal sensory afferents, to determine the effect on colonic pressure. We will compare the time required for the participant to complete their bowel emptying routine between a control period with digital rectal stimulation and a treatment period with electrical rectal stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Colasante-Garrido, MD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY; Dennis Bourbeau, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No